CLINICAL TRIAL: NCT05398874
Title: Clinical Efficacy of Ginkgo Biloba Extract in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Maryam Al-Haddad, Researcher, Kufa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC-13
Record Dates: First submitted 2022-05-20; First posted 2022-06-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginkgo + standard (Active Comparator): the patients received Ginkgo biloba extract in addition to standard treatment
  Interventions: Combination Product: Ginkgo biloba extract + standard treatment( paracetamol+Diclofenac100mg SR)
- placebo + standard (Placebo Comparator): the patients received a placebo in addition to the standard treatment
  Interventions: Combination Product: placebo in addition to the standard treatment

INTERVENTIONS:
Combination Product: Ginkgo biloba extract + standard treatment( paracetamol+Diclofenac100mg SR) — 120 mg leaf extract , twice daily in addition to Diclofenac 100 mg Once daily + paracetamol 1g Twice daily
  Other Names: Ginko Natrol company + Dolipran+Olfen 100 SR
  Arms: Ginkgo + standard
Combination Product: placebo in addition to the standard treatment — placebo in addition to the standard treatment
  Arms: placebo + standard

SUMMARY:
To assess the efficacy and safety of the Ginkgo biloba extract in patients with Knee OA.

ELIGIBILITY:
Inclusion Criteria:

* patients 40-75 years old with knee OA.
* Grade II and Grade III according to the Kellgrenn-Lawrence (KL) grading system of radiographic OA.

Exclusion Criteria:

* Pregnancy, breastfeeding
* Liver or renal problems
* Patient taking any drug that might interact with Ginkgo extract (eg. warfarin, etc.)
* patient with cardiovascular or cerebral vascular disorders, uncontrolled diabetes, allergic to ginkgo, recent surgery or hospital admission, >75 years old.
* Allergic or contraindicated to using NSAIDs

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
KOOS score | Changes occured : baseline , 2 weeks , 4 weeks ,and 8 weeks
  42 item questionnaire to assess pain, other symptoms, activities of daily living (ADL), sport and recreation function (Sport/Rec) and knee-related quality of life (QOL).

SECONDARY OUTCOMES:
IL-6 | Changes occured: baseline , 4 weeks,and 8 weeks
  Serum level of interleukin 6
TNF-alpha | Changes occured: baseline , 4 weeks,and 8 weeks
  Serum level of tumour necrosis factor - alpha
urinary CTX-II | Changes occured :baseline , 4 weeks,and 8 weeks
  C-terminal telopeptide of type II collagen from urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- Private Clinic, Najaf, N/A (Outside of US), Iraq

IPD SHARING:
Plan to Share IPD: Undecided